CLINICAL TRIAL: NCT07223164
Title: Validation of the Masimo Irregular Heartbeat Detection Algorithm in Participants Without Cardiovascular Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP-1102
Record Dates: First submitted 2025-10-29; First posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Specificity of Irregular Heartbeat Detection (Experimental): Specificity measure of performance of the Irregular Heartbeat Detection algorithm (evaluated for the finger and wrist form factors) against the Masimo Radius VSM® reference ECG. Each form factor will be evaluated independently of one another
  Interventions: Device: Masimo SET® and Masimo W1®

INTERVENTIONS:
Device: Masimo SET® and Masimo W1® — Pulse oximeter and wrist wearable device

SUMMARY:
Specificity measure of performance of the Irregular Heartbeat Detection algorithm (evaluated for the finger and wrist form factors) against the Masimo Radius VSM® reference ECG. Each form factor will be evaluated independently of one another

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 to 80 years of age.
* Comfortable to read and communicate in English.*
* Subject passes the health assessment conducted by qualified study personnel, confirming they are in adequate health to participate in the required procedures

  * This is to ensure the participant can provide informed consent and can comply with study procedures (as study material are currently available in English only).

Exclusion Criteria:

* Subject currently has a known cardiac disease condition.
* Subject is pregnant or breastfeeding.
* Subjects with a skin condition affecting the digits/chest, where the sensors are applied which would interfere with the path of lights (e.g., psoriasis, vitiligo, eczema, angioma, scar tissue, burn, fungal infection, substantial skin breakdown) or sensor adhesion.
* Skin condition which would preclude proper ECG placement.
* Subjects with nail polish or acrylic nails on the digits where sensor needs to be applied, who opt not to remove them.
* Subject is allergic to any supplies used in the study (e.g., ECG gel, adhesives).
* Subject has any medical condition which in the judgment of the investigator and/or study staff, renders them ineligible for participation in this study or subject is deemed ineligible by the discretion of the investigator/study staff.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Specificity of Masimo SET® | 1-2 hours
Specificity of Masimo W1® | 1-2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States